CLINICAL TRIAL: NCT04081259
Title: A Phase 1 Study of LY3214996, an ERK1/2 Inhibitor, in Patients With AML Who Are Not Candidates for Standard Therapy
Brief Title: LY3214996 in Patients With AML Who Are Not Candidates for Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Rahul Vedula, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-263
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; ERK; Relapsed; Refractory; LY3214996
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — LY3214996

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm B: Dose Escalation LY3214996 (Experimental): -LY3214996 will be administered by mouth once daily continuously throughout each treatment cycle for patients with inhibitors for fungal prophylaxis/treatment
  Interventions: Drug: LY3214996
- Arm A: Dose Expansion LY3214996 (Experimental): -LY3214996 will be administered by mouth once daily continuously throughout each treatment cycle for patients without inhibitors for fungal prophylaxis/treatment
  Interventions: Drug: LY3214996

INTERVENTIONS:
Drug: LY3214996 — LY3214996 is an extracellular signal-regulated kinase (ERK) inhibitor that is being developed as a treatment for patients with advanced cancer. ERK inhibitors stop the signal that a cancer cell receives telling it to grow.

SUMMARY:
This research study is evaluating a targeted therapy as a possible treatment for acute myeloid leukemia (AML) that has returned or not responded to standard treatment.

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is being studied.

The U.S. Food and Drug Administration (FDA) has not approved LY3214996 as a treatment for any disease.

LY3214996 is an extracellular signal-regulated kinase (ERK) inhibitor that is being developed as a treatment for patients with advanced cancer. ERK inhibitors stop the signal that a cancer cell receives telling it to grow. In this research study, the investigators are testing to see if LY3214996 is a safe treatment for AML that has returned or not responded to standard treatment. Several doses of the study drug will be explored in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed acute myeloid leukemia (AML) diagnosed per WHO criteria.
* Participants must have relapsed or refractory AML.
* Age ≥ 18 years.
* ECOG performance status ≤ 2
* Participants must have adequate organ function as defined below:

  * Direct Bilirubin ≤ 1.5 × institutional upper limit of normal (ULN)
  * AST (SGOT) and ALT(SGPT) ≤ 2.5 × institutional ULN, OR
  * AST (SGOT) and ALT (SGPT) ≤ 5 × institutional ULN if elevation is a result of leukemia
  * Creatinine Clearance ≥ 60 mL/min/1.73 m2 (calculated via the Cockcroft-Gault equation)
* The effects of LY3214996 on the developing human fetus are unknown. For this reason and because anti-cancer agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men and women treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of LY3214996 administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow and retain oral medication.
* Participants must have resolution of adverse events related to prior anti-cancer therapies to ≤ CTCAE Grade 2 or baseline
* Considerations of concurrent use of CYP3A4 inhibitors

Dose escalation phase:

* ARM A: Participants must not be receiving any concurrent antifungal agents that are moderate/strong CYP3A4 inhibitors. These include but are not limited to: isavuconazole, itraconazole, fluconazole, ketoconazole, posaconazole, and voriconazole.
* ARM B: Participants must be receiving concurrent antifungal agents that are moderate/strong CYP3A4 inhibitors. These include but are not limited to: isavuconazole, itraconazole, fluconazole, ketoconazole, posaconazole, and voriconazole.

Expansion Phase:

Participants not receiving concurrent antifungal agents that are moderate/strong CYP3A4 inhibitors are eligible to enroll at MTD determined upon completion of dose-escalation cohort Arm A. Participants receiving concurrent antifungal agents that are moderate/strong CYP3A4 inhibitors are eligible to enroll at MTD determined upon completion of dose-escalation cohort Arm B.

Exclusion Criteria:

* Participants who have had chemotherapy, other investigational therapy, immunotherapy, or radiotherapy within 2 weeks prior to the first dose of study medication. ATRA treatment is permitted with no required washout if treatment duration was for less than 1 week. Hydroxyurea is allowed with no required washout. For participants with an absolute peripheral blast count > 20 K/µL, hydroxyurea may be administered up to day 14 of protocol therapy with a maximum allowed dose of 6 g per day.
* Participants who have received oral tyrosine kinase inhibitors (TKIs) within 5 half-lives of the first dose of study medication.
* Participants who have had major surgery within 4 weeks prior to the first dose of study medication.
* Participants who have had a prior stem cell transplant (SCT) within 90 days prior to the first dose of study medication. Additionally, participants having undergone prior SCT must be off calcineurin inhibitor therapy for at least 28 days prior to the first dose of study medication.
* Participants with active > Grade 1 acute or chronic Graft v. Host Disease (GvHD) who are receiving immunosuppressive therapy other than prednisone. Use of prednisone is permitted only if participants have been maintained at a steady dose of < 20 mg/day for at least 5 days prior to the first dose of study medication.
* Participants with known active CNS leukemia involvement. Participants with no known history of CNS leukemia are not required to undergo lumbar puncture (LP) for trial eligibility unless the participant is symptomatic as judged by the treating investigator. Participants with a history of CNS leukemia involvement are eligible provided that the CNS disease has been adequately treated and cleared prior to study enrollment as judged by the treating investigator.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to LY3214996.
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because LY3214996 is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with LY3214996, breastfeeding should be discontinued if the mother is treated with LY3214996. A negative serum pregnancy test is required for women of childbearing potential prior to study entry.
* Participants who are known to be seropositive for human immunodeficiency virus (HIV) or hepatitis B or C. Testing is not required for eligibility.
* Participants with a history or findings of central or branch retinal artery or venous occlusion with significant vision less, or other retinal diseases causing visual impairment as determined by an ophthalmologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-26 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 21 days
  Toxicities occurring following administration of protocol therapy, measured using CTCAE 5.0 criteria.

SECONDARY OUTCOMES:
Overall Response Rate | 6 months
  Rate of complete remission (CR), CR with incomplete count recovery (CRi), and partial remission (PR) using IWG and ELN criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Vedula, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to the sponsor. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu